CLINICAL TRIAL: NCT06666998
Title: Real-World Pharmacokinetic/Pharmacodynamic Study of Eravacycline in Critically III Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Lingai Pan, Associate Clinical Professor, Sichuan Provincial People's Hospital
Other Study IDs: LPan2
Record Dates: First submitted 2024-10-25; First posted 2024-10-31 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Eravacycline; Pharmacokinetics; Bacteria Infection; Bacterial Resistance to Antimicrobial; Empirical Antimicrobial Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this study is to evaluate the efficacy of Eravacycline in the treatment of patients with bacterial infection and to assess the pharmacokinetics of Eravacycline and to establish a population pharmacokinetic model of Eravacycline.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female aged 18-75 years
* Not respond to initial empirical treatment, treatment time to reach Eravacycline steady-state concentration
* Empirical antimicrobial treatment is ineffective
* Eravacycline application for ≥ 3 days
* Understand and sign informed consent

Exclusion Criteria:

* Urinary tract infection
* Allergic to Eravacycline, Tigecycline antibiotics or any excipients or have previously experienced serious adverse reactions
* Any unstable or potentially endangering the safety of the subject and their compliance with the study as judged by the investigator; comorbidities or social circumstances that can make the subject unable to follow the study plan or even endanger the safety of the patient
* Patients expected to survive for no longer than 48h.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 critically infected patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Clinical remission rate | At the end of treatment；2 weeks（estimated）
  Completion of scheduled course of treatment; ≤14 days of treatment; treatment not restarted within 48 hours of discontinuation
Microbiological efficacy | From enrollment to the end of treatment at 28 days
  Evaluate at the end of treatment and at post-treatment (discharge) in patients who met all clinical evaluation criteria and who had positive bacteriologic cultures prior to treatment, and bacterial clearance was calculated using the results of post-treatment follow-up (discharge) as the primary endpoint of evaluation.Performing safety observation (including coagulation dysfunction and other adverse reactions)

SECONDARY OUTCOMES:
Develop Population Pharmacokinetic Model | From enrollment to the end of treatment at 28 days
  Initial testing perform at first dose and steady-state testing perform at the seventh dose.Calculation of all-eravacycline fAUC using the linear trapezoidal method.Multiple regression analysis use to generate the best model equation for estimating the fAUC using the concentration of eravacycline at each sampling point in the modeling group as the independent variable and the fAUC as the dependent variable.

IPD SHARING:
Plan to Share IPD: Undecided